CLINICAL TRIAL: NCT03409640
Title: The Rate of Symptomatic and Asymptomatic Non-malignant, Non-infective Soft Tissue Masses in Primary Metal on Metal Hip Replacement.
Brief Title: Metal-on-metal Hip Replacement MRI Study
Status: Completed | Type: Observational
Sponsor: Zimmer Biomet (Industry)
Responsible Party: Sponsor
Other Study IDs: ORTHO.CR.GH34
Record Dates: First submitted 2018-01-08; First posted 2018-01-24 (Actual); Last update posted 2018-01-24 (Actual); Status verified 2018-01

CONDITIONS: Hip Athroplasty Using M2a Magnum

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is being conducted to determine the rate of symptomatic and asymptomatic nonmalignant, noninfective soft tissue mass presence (referred to in the literature as pseudotumour, ALVAL, ARMD, cysts or lesions) in primary metal on metal hip replacement patients. The primary objective of the study is to determine the prevalence of masses in unbiased Metal on Metal (MoM) samples drawn from one study centre. The subjects receiving the Metal on Metal devices will be observed at two specific time points. Secondary objectives are to evaluate whether the occurrence of masses is related to any of several potential factors including patient and implant characteristics and time since the implant procedure took place.

ELIGIBILITY:
Inclusion Criteria:

• Patients implanted with the M2a Magnum who were evaluated via MRI and metal ion analysis between 2012 and 2013.

Exclusion Criteria:

* If the primary device was implanted for less than 36 months (in the case of patients already revised) or has been in place for less than 36 months (in the case of patients with the device still in place).
* If the patient is contraindicated for any of the diagnostic tests.
* If the patient fails to consent to participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving either the M2a Magnum or M2a 38mm Metal on Metal primary hip replacement devices from a single study centre.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-01-17 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
MRI Scoring change in soft tissue mass size | 36 months after primary device implantation
  MRI Score - monitor number and size of soft tissue lesions

SECONDARY OUTCOMES:
Radiographic assessment | 36 months after primary device implantation
  Assess acetabular cup inclincation and version
Oxford Hip Score | 36 months after primary device implantation
  Oxford Hip Score, score range 0 (worst) to 48 (best)
UCLA Activity Score | 36 months after primary device implantation
  UCLA activity scale, range: 1 defined as "no physical activity, dependent on others" to 10 defined as "regular participation in impact sports."
EQ-5D | 36 months after primary device implantation
  EQ-5D Index score; Patient Reported Outcome
Metal Ion Levels | 36 months after primary device implantation
  Chromium and Cobalt metal ion levels in blood

CONTACTS AND LOCATIONS:
Locations (1):
- Basingstoke and North Hampshire Hospital, Basingstoke, United Kingdom